CLINICAL TRIAL: NCT00002454
Title: Phase II Study of Immunotherapy With Autogenous Papilloma Vaccine in Patients With Recurrent Juvenile Papilloma of the Larynx
Brief Title: Papilloma Virus Vaccine Therapy in Treating Young Patients With Recurrent Papilloma of the Larynx
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000071657; NJ-LAR-1; NJ-M-41-1976
Record Dates: First submitted 1999-11-01; First posted 2004-02-27 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2002-01

CONDITIONS: Precancerous Condition
Keywords: lung papilloma
MeSH Terms: conditions — Precancerous Conditions | interventions — FANG vaccine

INTERVENTIONS:
Biological: autologous tumor cell vaccine

SUMMARY:
RATIONALE: Vaccines made from papilloma virus cells may make the body build an immune response to and kill papilloma cells.

PURPOSE: Phase II trial to study the effectiveness of papilloma virus vaccine in treating young patients with recurrent papilloma of the larynx.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the immune response in patients with juvenile papilloma of the larynx treated with autogenous vaccine derived from each patient's own tumor.

OUTLINE: Patients receive autogenous papilloma vaccine intradermally and subcutaneously weekly for 20 weeks.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of severe recurrent juvenile papilloma of the larynx requiring surgery at least 4 times per year Condition must have existed for more than 1 year

PATIENT CHARACTERISTICS: Age: 1 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1971-12

CONTACTS AND LOCATIONS:
Overall Officials: James M. Oleske, MD, Study Chair — Rutgers, The State University of New Jersey
Locations (1):
- New Jersey Medical School, Newark, New Jersey, United States

REFERENCES:
- [Result] Oleske J, Fishman D, Cooper R, et al.: Autogenous vaccine in the treatment of laryngeal papilloma. In: Proceeding of the 12th International Congress of Chemotherapy, 1981. pp 1099-1101.
- [Result] Oleske JM, Kushnick T. Juvenile papilloma of the larynx. Am J Dis Child. 1971 May;121(5):417-9. doi: 10.1001/archpedi.1971.02100160087011. No abstract available. PMID 4326367